CLINICAL TRIAL: NCT03131310
Title: Managment of Cardiorespiratory Arrest
Acronym: clinicalaudit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fefe Saad, Doctor, Assiut University
Other Study IDs: Assiut university117100107
Record Dates: First submitted 2017-04-23; First posted 2017-04-27 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Assess the Quality Ofmanagement of Children With Cardiorespiratory Arrest in Assuit University Children Hospital According to the( A H A)Guidelines
MeSH Terms: interventions — Clinical Audit

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: clinical audit — is to assess the quality of care and management of children with cardiorespiratory arrest admitted to assuit university children hospital according to the American Heart Association (AHA) Guidelines for Cardiopulmonary Resuscitation

SUMMARY:
CPR will be done based on American Heart Association Guidelines for Cardiopulmonary Resuscitation (2015) and Emergency Cardiovascular Care of Pediatric and Neonatal Patients.

DETAILED DESCRIPTION:
the present study is to assess the quality of care and management of children with cardiorespiratory arrest admitted to assuit university children hospital according to the American Heart Association Guidelines for Cardiopulmonary Resuscitation (2015) and Emergency Cardiovascular Care of Pediatric and Neonatal Patients searching for defect,obstacles,or need to improve health service.

CPR will be done based on American Heart Association Guidelines for Cardiopulmonary Resuscitation (2015) and Emergency Cardiovascular Care of Pediatric and Neonatal Patients.

ELIGIBILITY:
Inclusion Criteria:

* Seriously ill Patients who will be admitted with or will be developed cardiorespiratory arrest and undergo CPR.

Age2 month to 18 years. Both sex.

Exclusion Criteria:

* Traumatic cause (blunt, penetrating, burn) of arrest

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: the present study is to assess the quality of care and management of children with cardiorespiratory arrest admitted to assuit university children hospital according to the American Heart Association (AHA) Guidelines for Cardiopulmonary Resuscitation (CPR) (2015) and Emergency Cardiovascular Care (ECC) of Pediatric and Neonatal Patients searching for defect,obstacles,or need to improve health service. CPR will be done based on American Heart Association (AHA) Guidelines for Cardiopulmonary Resuscitation (CPR) (2015) and Emergency Cardiovascular Care (ECC) of Pediatric and Neonatal Patients.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
managment of cardiorespiratory arrest in children | one year
  assesment of cardiorespiratory ressucitation

IPD SHARING:
Plan to Share IPD: Undecided
assess the quality of care and management of children with cardiorespiratory arrest admitted to assuit university children hospital according to the American Heart Association (AHA) Guidelines for Cardiopulmonary Resuscitation